CLINICAL TRIAL: NCT05274568
Title: Proof of Mechanism Study to Evaluate Binding of Alfa-synuclein by [18F]UCB-2897 in Participants With Parkinson's Disease or Multi-system Atrophy
Brief Title: Proof of Mechanism Study to Evaluate Binding of Alfa-synuclein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10616
Record Dates: First submitted 2022-02-01; First posted 2022-03-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Multisystem Atrophy; Healthy Volunteer
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]UCB-2897 (Experimental): Administration of Investigational Agent:
  Study center personnel will administer [18F]UCB-2897 as an IV injection. Prior to PET imaging, participants will have an IV catheter (for radiopharmaceutical administration) inserted according to standard clinical practice. Each participant will receive a single injection of [18F]UCB-2897. [18F]UCB-2897 will be injected IV at a dose of not more than 10 mCi, with a maximum mass dose of 10 μg and maximum volume of 10 mL. The injection will be followed by a 10 mL saline flush. Qualified study staff will accompany participants during PET imaging procedures.
  Interventions: Drug: [18F]UCB-2897

INTERVENTIONS:
Drug: [18F]UCB-2897 — Investigational Agent:
  [18F]UCB2897 is a clear solution formulated for intravenous (IV) injection. The product [18F]UCB2897is delivered in normal saline (0.9 % sodium chloride [NaCl]) formulated with the intent to contain approximately 3.3 % (v/v) ethanol (EtOH), polysorbate-80 (PS-80, 3.73 μL/mL) and sodium ascorbate (4.67 mg/mL). The final product bears a label with the following items: total activity (mCi), volume (mL), strength (mCi/mL), calibration date and time, batch number, and shelf life. [18F]UCB2897 will be stored at ambient temperature in its original container.

SUMMARY:
The overall goal of this protocol is to:

Evaluate [18F]UCB-2897 as an α-synuclein targeted radiopharmaceutical.

The primary objective is:

• Confirm a specific α -synuclein signal with [18F]UCB-2897 in participants with PD and/or MSA relative to healthy volunteers

Secondary and exploratory objectives are:

* Determine the safety and tolerability of microdose [18F]UCB-2897
* Evaluate preliminary dosimetry of [18F]UCB-2897

Additional exploratory objectives are:

* Determine the pharmacokinetics / metabolism of [18F]UCB-2897
* Determine the optimal imaging protocol for [18F]UCB-2897

DETAILED DESCRIPTION:
This is a first in human [FiH], open-label study to assess the imaging characteristics, kinetics, and safety of [18F]UCB-2897 in participants with MSA, participants with PD, and healthy participants. Up to 2 participants with MSA, up to 8 participants with PD, and up to 5 healthy volunteers will be enrolled from the available database at Invicro, through advertising, and through physician referral. Participants will be enrolled in 2 parts that may be run concurrently: Part A (up to 2 participants with PD and up to 2 participants with MSA) and Part B (up to 6 participants with PD and up to 5 healthy volunteers). Data will be reviewed on an ongoing basis throughout the study, at least at the end of Part A.

All participants will attend the following (with exceptions noted):

* Screening
* [18F]UCB-2897 positron emission tomography (PET) Imaging Visit (including brain PET imaging or whole-body PET imaging)
* Follow-up Phone Call
* Amyloid PET Imaging Visit (not performed for all participants)
* DaTscan single photon emission computed tomography (SPECT) Imaging Visit (not performed for all participants)

During Screening, participants will undergo assessments to confirm study eligibility, including an MRI scan (unless a previously acquired approved scan is available) for participants who will have brain PET imaging. Participants with MSA and PD will also have a DaTscan SPECT scan during Screening (unless a previously acquired approved scan is available).

Within 4 weeks of the start of Screening, participants will attend a [18F]UCB-2897 PET Imaging Visit. Participants with MSA, participants with PD, and up to 2 healthy volunteers will undergo brain PET imaging, including one injection of [18F]UCB-2897, one brain PET scan lasting up to 2 hours, and arterial blood sampling. If the participant does not consent to arterial blood sampling or the study team deems it appropriate based on emerging data, venous blood samples may be collected in lieu of arterial blood samples. Brain PET imaging and blood data will be used to assess α-synuclein binding by [18F]UCB-2897. Up to 3 healthy volunteers will undergo whole-body PET imaging assessments, including one injection of [18F]UCB-2897, a series of whole-body PET scans lasting up to 6 hours, and urine collection. Whole-body PET imaging and urine samples will be assessed for a preliminary evaluation of [18F]UCB-2897 dosimetry. During PET imaging (both brain and whole-body), safety assessments will be performed to evaluate the safety and tolerability of [18F]UCB-2897, including ECGs, physical and neurological examinations, clinical laboratory samples, and vital sign measurements.

A Follow-up Phone Call to the participant will be conducted 4 days (± 2 days) post-injection of [18F]UCB-2897 to confirm participant well-being and to collect information about any new adverse events (AEs).

If the study team considers that further investigation on potential cross-binding with beta (β)-amyloid is needed, participants with MSA or PD will attend an Amyloid PET Imaging Visit and have amyloid PET imaging performed with an approved amyloid tracer (unless a previously acquired approved scan is available). Additionally, if needed for further interpretation of data, healthy volunteers who received brain PET imaging may have a DaTscan SPECT scan (unless a previously acquired approved scan is available).

When the participant completes his or her final study visit, the participant will be formally released from the study.

ELIGIBILITY:
Inclusion Criteria for all Participants:

* Participant is able to provide informed consent, which must be obtained before any study procedures are performed.
* Female participants must not be of childbearing potential, or if they are of childbearing potential must agree to use contraception and not donate eggs.

  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (ie, removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the principal investigator (PI) (eg, Müllerian agenesis).
  * Women of childbearing potential must commit to remain abstinent (refrain from heterosexual intercourse) or use 2 forms of birth control, 1 of which is a barrier contraception method, for the duration of the study and 30 days after study completion. Periodic abstinence (eg, calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
  * Women of childbearing potential must commit to not donate ova for the duration of the study and 30 days after study completion.
* Male participants with partners of childbearing potential must commit to the use of 2 methods of contraception, 1 of which is a barrier method for male participants for the study duration and 90 days after study completion.
* Male participants must not donate sperm for the study duration and for 90 days after study completion.
* Willing and able to cooperate with study procedures.
* For participants who will have arterial cannulation performed, adequate circulation to the hand for safe placement of arterial line (as determined by Allen's test) and blood clotting (Prothrombin Time [PT] and Partial Thromboplastin Time [PTT]).
* If participant takes bupropion, participant must agree to hold this medication for at least 12 hours prior to DaTscan imaging (if performed).
* OTC medication (except acetaminophen), herbal supplements, dietary supplements, or vitamins approved by the Investigator, must be stable within 2 weeks prior to initial dosing.

Additional inclusion criteria for participants with MSA:

* Males and females aged ≥ 50 years.
* Diagnosis of probable MSA, according to Consensus Clinical Diagnostic Criteria for MSA and a consistent MRI scan performed either at Screening or previously acquired.
* Evidence of dopamine transporter (DaT) deficit on DaTscan performed either as part of Screening or previously acquired.
* Medications taken for symptomatic treatment must be maintained on a stable dosage regimen for at least 30 days before Screening Visit.
* Ability to tolerate lying in the scanner for up to 2 hours, without excessive head or jaw tremor or dyskinesia sufficient to cause significant motion artifact on the PET scans.
* Prescription drugs approved by the Investigator must be stable within 4 weeks prior to initial dosing.

Additional inclusion criteria for participants with PD:

* Males and females aged ≥ 50 years.
* Clinical diagnosis of PD (early, moderate, or severe) for > 6 years, according to medical history, and L-DOPA responsive.
* Evidence of DaT deficit on DaTscan performed either as part of Screening or previously acquired.
* Medications taken for symptomatic treatment must be maintained on a stable dosage regimen for at least 30 days before Screening Visit.
* Ability to tolerate lying in the scanner for up to 2 hours, without excessive head or jaw tremor or dyskinesia sufficient to cause significant motion artifact on the PET scans.
* Prescription drugs approved by the Investigator must be stable within 4 weeks prior to initial dosing.

Additional inclusion criteria for healthy volunteers:

* Males and females aged ≥18 years.
* Healthy with no clinically relevant finding on physical examination at Screening.
* No family history of α-synucleinopathy, including PD or other early-onset neurological disease associated with dementia.
* No personal history of clinically significant neurologic and/or psychiatric disorders.
* No cognitive impairment as judged by the Investigator.

Exclusion Criteria for all participants:

* Pregnant, lactating or breastfeeding.
* Current or prior history of any alcohol or drug abuse in the past 2 years to be verified by urine drug screen.
* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
* History of immunodeficiency diseases, including a positive HIV test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody test result.
* Known history of hypersensitivity, including hypersensitivity to the active substances used for DaTscan, [18F]UCB2897, and/or [18F]florbetapir or derivatives, or to any of the associated excipients.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* Are claustrophobic or otherwise unable to tolerate the imaging procedure.
* MRI with clinically significant structural abnormalities, other than those expected for MSA or PD for those participants.
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, central nervous system (CNS) aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.
* Participant has received an investigational drug within 30 days or five half-lives prior to Day 1, whichever is longer.
* Participant has received treatment with a drug, antibody or vaccine targeting α-synuclein.
* Prior participation in other research protocols, clinical care, or occupational exposure during the past year that would result in radiation exposure to an effective radiation dose exceeding the acceptable annual limit established by the US Federal Guidelines (effective dose of 50 mSv, including the procedures in this clinical protocol).
* For participants receiving DaTscan imaging, ongoing treatment with methylphenidate, modafinil, metoclopramide, alpha methyldopa, reserpine, or amphetamine derivative is prohibited 24 hours or during a period corresponding to 5 half-lives of the compound, whichever longer, prior to DaTscan imaging.

For participants who will have arterial blood sampling, treatment with any antihemostasis medication (eg, warfarin, heparin, thrombin inhibitors, Factor Xa inhibitors, streptokinase, urokinase, tissue plasminogen activators) within 2 weeks of the planned arterial cannula placement.

• Participant is, in the opinion of the Investigator, unsuitable in any other way to participate in this study.

Additional exclusion criteria for healthy volunteers:

* BMI < 16 or > 35.
* The participant is currently exposed to nicotine products or had regular nicotine exposure within a six-month period, to be verified by urine cotinine screening.
* Use of any prescription drugs (except approved forms of birth control) or herbal supplements, within 4 weeks prior to Screening.

Additional exclusion criteria for participants with MSA:

• Evidence of early frequent falls or eye movement abnormalities consistent with progressive supranuclear palsy (PSP).

Additional exclusion criteria for participants with PD:

* The participant is currently exposed to nicotine products or had regular nicotine exposure within a six-month period, to be verified by urine cotinine screening.
* Evidence of early frequent falls or eye movement abnormalities consistent with PSP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Quantitative analysis of [18F]UCB-2897 brain PET scans | Day 1: PET Imaging Visit
  [18F]UCB-2897 uptake and kinetics will be examined in the MSA, PD, and healthy volunteer groups descriptively and quantitatively to describe the α-synuclein deposition as measured by [18F]UCB-2897 across multiple brain regions.
Whole-body Biodistribution Outcome Measures | [18F]UCB-2897 PET Imaging Visit
  For whole-body biodistribution, total source organ counts over time based on an individualized VOI template will be used to determine radiation absorbed dose estimates and whole-body effective doses based on the MIRD methodology.
Safety Outcome Measures | Screening, pre-injection, and at the completion of imaging
  Safety will be evaluated throughout the study. Safety will be evaluated by assessing incidence and severity of AEs, results from measurements of vital signs and ECGs, results from measurements for parameters of hematology, clinical chemistry, and urinalysis.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, MD, Ph.D, Principal Investigator — Principal Investigator; Joyce Gibbons, PA-C, Principal Investigator — Sub-Investigator; Amy Knorr, MD, Principal Investigator — Sub-Investigator
Locations (1):
- Invicro, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://invicro.com/